CLINICAL TRIAL: NCT05337449
Title: Evaluation Of Changes in Children's Oral Health-Related Quality of Life Following Treatment of Early Childhood Caries With Caries Arrest Technique Using Silver Diamine Fluoride Versus Conventional Drill and Fill Technique A Randomized Clinical Trial
Brief Title: Oral Health-Related Quality of Life of Early Childhood Caries Using Silver Diamine Fluoride Versus Drill and Fill Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gala Sharif Osman, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHrQL in ECC treated with SDF
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-04

CONDITIONS: Oral Health Related Quality of Life; Early Childhood Caries
MeSH Terms: interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: for both the intervention group and control group, the procedure and follow up will be done parallel to each other
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- silver diamine fluoride (Active Comparator)
  Interventions: Other: silver diamine fluoride; Other: conventional composite resin restoration
- conventional composite resin restoration (Active Comparator)
  Interventions: Other: silver diamine fluoride; Other: conventional composite resin restoration

INTERVENTIONS:
Other: silver diamine fluoride — silver diamine fluoride is a colorless with high PH topical fluoride solution of 38% weight/volume use for arresting early childhood caries
Other: conventional composite resin restoration — Dental composite resins are dental cement made of synthetic resins which were insoluble, of good tooth-like appearance, insensitive to dehydration, and easy to manipulate.

SUMMARY:
The clinical trial aims to compare children's oral health-related quality of life (OHrQL) following caries arrest technique using SDF versus conventional drill and fill in the children with ECC

DETAILED DESCRIPTION:
Early childhood caries (ECC) has been an increasing issue in many countries and has become a significant health problem, especially in socially disadvantaged populations. ECC is a specific form of caries that occurs in children with primary teeth. ECC is characterized as "the early onset of caries in young children with often fast progression which can finally result in complete destruction of the primary dentition".

Management of cavitated carious lesions in primary teeth in very young children is time-consuming due to their lack of cooperation, so one of the alternative procedures could be performed with silver diamine fluoride (SDF), to its effectiveness in arresting the activity of carious lesions (cavitated and non-cavitated). It is easy to apply even outside dental offices, and relatively inexpensive solutions can be used particularly when compared to restorative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children Aged 3 to 5 years, in good general health and medically within normal.
* The parents provided written informed consent.
* Carious vital primary molars with reversible pulpitis.
* Restorable teeth.
* Normal Radiographic findings.

Exclusion Criteria:

* Unable to attend follow-up visits.
* Refusal of participation.
* Previously accessed teeth.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Oral Health to Quality of Life | 6 month intervene
  will be evaluated by a questioner answered by the parents

SECONDARY OUTCOMES:
The cost effectiveness | 6 month intervene
  will be measured using ICER (incremental cost-effectiveness ratio)
Parental satisfaction | 6 month intervene
  will be measured by Direct questioning to the parents.
Side effects | 6 month intervene
  will be measured by Direct questioning to the parents.
Time of the procedure | 6 month intervene
  will be measured by stopwatch
Postoperative pain and sensitivity | 6 month intervene
  will be measured by Visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Gala Osman, BDS, Principal Investigator — Cairo University; Sherine Younes, Professor, Study Director — Cairo University; Passant Nagii, PHD, Study Director — Cairo University